CLINICAL TRIAL: NCT00312520
Title: The Efficacy and Safety of Intravenous Pulse Steroids Compared to Standard Oral Steroids in the Treatment of Problematic Hemangiomas in Infants: A Randomized Controlled Trial
Brief Title: Pulse Steroids Versus Oral Steroids in Problematic Hemangiomas of Infancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Society for Pediatric Dermatology (Other)
Responsible Party: Principal Investigator, Elena Pope, Head, Section of Dermatology, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0020020166
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Hemangiomas
MeSH Terms: conditions — Hemangioma | interventions — Prednisolone; Methylprednisolone

INTERVENTIONS:
Drug: prednisolone
Drug: methylprednisolone

SUMMARY:
The purpose of the study is to determine if pulse steroids are more efficacious and safer than the standard treatment with oral corticosteroids.

DETAILED DESCRIPTION:
Currently there is no prospective study in hemangioma patients answering critical questions such as: which type of steroid should be used,how much should we use and for how long. This study is an investigator blinded study with two arms:one arm is receiving standard treatment with daily oral corticosteroids and the other is receiving intravenous pulse corticosteroids daily for 3 days, monthly for 3 months. The main outcome of the study is assess the efficacy of each treament modality as the percentage improvement in the hemangioma's appearance. The secondary outcomes are the safety profiles of the two drugs and the changes in the angiogenesis markers as a result of treatment intervention.

ELIGIBILITY:
Inclusion Criteria:

* problematic facial hemangiomas (periorbital/facial hemangiomas with potential visual obstruction, large/dysfiguring hemangiomas)
* 1-4 months of age
* signed consent form

Exclusion Criteria:

* refusal to participate
* age > 4 months
* complicated nonvisible hemangiomas
* congenital heart disease

Ages: 1 Month to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Start 2002-07 (Actual); Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Percent improvement in the appearance of hemangioma

SECONDARY OUTCOMES:
Frequency of side-effects experienced by the patients
Changes in the angiogenesis markers

CONTACTS AND LOCATIONS:
Overall Officials: Elena Pope, MD, Msc, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada